CLINICAL TRIAL: NCT07015021
Title: The Efficacy and Safety of the Combination Therapy of Daratumumab, Cabozantinib, Pomalidomide, and Dexamethasone (D-KPd) in the Treatment of High-risk First-time Relapsed or Primary Refractory MM Patients: a Randomized, Open Label, Single Arm, Single Center Clinical Study
Brief Title: The Efficacy and Safety of the Combination Therapy of Daratumumab, Cabozantinib, Pomalidomide, and Dexamethasone (D-KPd) in the Treatment of High-risk First-time Relapsed or Primary Refractory MM Patients
Acronym: DKPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Fu chengcheng PhD, Deputy Director, Department of Hematology, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKPD-MM01
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; Carfilzomib; Daratumumab; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk First-time Relapsed or Primary Refractory MM Patients (Experimental): Daratumumab: 16mg/Kg, IV or 1800mg Sc; C1-2 d1,8,15,22; C3-6 d1,15; C7-12 d1。 Cafizomide: 20mg/m2; C1-8 d1,2,8,9,15,16； C9-12 d1,2,15,16； After tolerance to 20mg/m2, the dose of C1D1 and C1D2 can be adjusted to 27g/m2.
  Pomalidomide: 4mg, PO,d1-21。 Dexamethasone: 20mg, po,d1, 2,8,9,15,16,22,23.
  Interventions: Drug: Daratumumab; Drug: Cafizomide; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab: 16mg/Kg, IV or 1800mg Sc; C1-2 d1,8,15,22; C3-6 d1,15; C7-12 d1
Drug: Cafizomide — Cafizomide: 20mg/m2; C1-8 d1,2,8,9,15,16； C9-12 d1,2,15,16；After tolerance to 20mg/m2, the dose of C1D1 and C1D2 can be adjusted to 27g/m2.
Drug: Pomalidomide — Pomalidomide: 4mg, PO,d1-21
Drug: Dexamethasone — Dexamethasone: 20mg, po,d1, 2,8,9,15,16,22,23.

SUMMARY:
This study is a prospective, single center, single arm phase II clinical trial. The study population consists of patients who have received treatment with VRd or VRd lite regimens for 2-8 courses in the past and have achieved therapeutic effects, but have progressed during treatment (primary refractory), experienced clinical recurrence for the first time after treatment, or progressed or recurred after the first transplant (without entering maintenance therapy). 72 patients are planned to be enrolled and receive 4 courses of induction therapy with D-KPd regimen for the first efficacy evaluation. For patients with ≥ SD, if the patient has ≥ PR and is suitable for ASCT, ASCT treatment will be given. For patients with<PR or not suitable for ASCT, 4 courses of consolidation therapy with D-KPd regimen will be continued for the second efficacy evaluation SD patients continue to receive 4 courses of D-KPd regimen consolidation treatment. D-KPd dosing regimen: Daratumumab: 16mg/Kg, IV or 1800mg Sc; C1-2 d1,8,15,22; C3-6 d1,15; C7-12 d1。 Cafizomide: 20mg/m2; C1-8 d1,2,8,9,15,16； C9-12 d1,2,15,16； After tolerance to 20mg/m2, the dose of C1D1 and C1D2 can be adjusted to 27g/m2. Pomalidomide: 4mg, PO,d1-21。 Dexamethasone: 20mg, po,d1, 2,8,9,15,16,22,23. If the age is over 75 years old, the Dex dose is halved. The main efficacy endpoint after 12 treatment courses is: ORR； Secondary efficacy endpoint indicators: mPFS, mOS, ≥ VGPR rate, MRD negative rate, safety

DETAILED DESCRIPTION:
Considering that the majority of initial treatment patients in China have already received pre-treatment with lenalidomide and bortezomib, the vast majority of patients who experience disease progression will be refractory to lenalidomide and exposed to bortezomib. Both carfilzomib and pomalidomide have been shown to be effective against lenalidomide resistance, and the combination of carfilzomib, pomalidomide, and dexamethasone has a combined anti myeloma effect. Currently, the combination of the three drugs has become a routine treatment for RRMM patients. Previous studies abroad have shown that the D-KPd regimen combined with four drugs can prolong the median PFS of RRMM patients (with a median prior treatment line of 2) to 30.9 months. Another study led by the University of Chicago showed that for patients with first-time recurrent RRMM, the D-KPd regimen had longer mPFS and mOS compared to the KPd regimen. However, there are currently no relevant reports on the efficacy data of D-KPD regimen in China. Considering regional and ethnic differences, as well as the lack of particularly good treatment options for high-risk first-time relapse and primary refractory MM patients in China, we plan to design this prospective, single center, single arm clinical trial to determine the effectiveness and safety of D-KPd regimen for high-risk first-time relapse or primary refractory MM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 18 years old;
2. Functional high-risk patients: Patients who have previously received treatment with VRd or VRd lite regimens for 2-8 courses and achieved therapeutic effects, but have progressed during treatment (primary refractory), experienced clinical recurrence for the first time after treatment, or developed progression or recurrence after the first transplantation (not entered maintenance treatment).
3. Multiple myeloma patients with measurable M protein must meet at least one of the following three criteria: 1) serum M protein ≥ 10 g/L; 2) Urinary M-protein ≥ 200 mg/24h; 3) In the case of abnormal serum free light chain ratio, the affected free light chain level is ≥ 100 mg/L [18];
4. Physical condition (ECOG) score 0-2 points, expected survival period ≥ 3 months;
5. Hematology meets the following conditions: ANC ≥ 1.0 × 109/L (G-CSF is not allowed to be used within 14 days after screening), patients with ANC<1.0 × 109/L can consider screening based on specific circumstances and additional monitoring after discussing with PI and obtaining PI approval; When the number of myeloma cells is less than 50%, PLT ≥ 75 × 109/L, and when the number of myeloma cells is ≥ 50%, PLT ≥ 50 × 109/L (platelet transfusion is not allowed within 7 days after screening); Hemoglobin level ≥ 7.5g/dL.
6. The creatinine clearance rate measured or calculated by the patient is ≥ 30mL/min.
7. The liver, heart and other major organs meet the requirements of the following laboratory examination indicators (conducted within 7 days before treatment):

1) Total bilirubin ≤ 1.5 times the upper limit of normal value (for the same age group); 2) Aspartate transaminase (AST) and alanine aminotransferase (ALT) are ≤ 2.5 times the upper limit of normal values for the same age group; 3) Myocardial enzymes are less than twice the upper limit of normal values for the same age group; 4) The ejection fraction measured by echocardiography (ECHO) is within the normal range.

8. Women of childbearing age (FCBP) subjects must have a negative serum pregnancy test 21 days prior to enrollment and agree to use an effective contraceptive method during all study drug periods and within 30 days after the last receipt of the study drug (if pregnancy tests may be conducted more frequently according to local guidelines). This protocol defines FCBP as sexually mature women who have not undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, or have not experienced natural menopause for at least 24 consecutive months (i.e. have had menstruation at any time during the past 24 consecutive months); If there is sexual activity with FCBP, male participants must use an effective barrier contraceptive method during the study period and within 3 months after the last receipt of the study drug. Male participants are not allowed to donate sperm during the treatment period and within 90 days after receiving the study drug for the last time. Male participants whose partners are pregnant must abstain from sexual activity or use condoms during vaginal intercourse; 10. Clearly understand the content of the experiment, voluntarily participate and complete the experiment, and sign the informed consent form. The informed consent form shall be signed by the patient or their immediate family members. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, an informed consent form shall be signed by the legal guardian or the patient's immediate family members; 11. It is necessary to agree to comply with all research requirements, follow-up schedules, outpatient treatment, necessary concomitant medication therapy, and laboratory monitoring.

Exclusion Criteria:

1. Non active multiple myeloma, including MGUS and smoking myeloma;
2. Subjects with POEMS syndrome or known/suspected amyloidosis in any organ;
3. Subjects with plasma cell leukemia: patients with a proportion of peripheral plasma cells ≥ 5% and/or an absolute value of peripheral plasma cells ≥ 0.5 × 109/L;
4. Patients who have been exposed to daratumumab in the past;
5. Previous malignant tumors that require treatment or have evidence of recurrence within the 5-year period prior to the first study medication [excluding basal cell carcinoma of the skin and the following in situ cancers: squamous cell carcinoma, bladder in situ carcinoma, endometrial in situ carcinoma, cervical in situ carcinoma/atypical hyperplasia, prostate cancer incidentally discovered histologically (TNM staging T1a or T1b), or breast in situ carcinoma];
6. Hepatitis B serum positivity (defined as positive detection of hepatitis B surface antigen [HBsAg]). The subjects whose infection has subsided (that is, the subjects whose HBsAg is negative but whose hepatitis B B core antigen antibody [anti HBc] and/or hepatitis B B surface antigen antibody [anti HBs] are positive) must use real-time polymerase chain reaction (PCR) to detect the level of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) for screening. PCR positive individuals will be excluded. Exception: Serological results indicate HBV vaccination (with anti HBs positivity as the sole serological marker) and subjects with a known history of HBV vaccination do not require PCR detection of HBV DNA;
7. Known to be HIV positive;
8. Uncontrolled active infections, or acute active infections, require systemic use of antibiotics, antiviral drugs, or antifungal drugs within two weeks prior to the first use of medication;
9. History of VTE or cerebral infarction before treatment;
10. The patient has uncontrolled or severe cardiovascular disease, including hypertension that has not been effectively controlled within the past 6 months (hypertension is defined as: non same day 3 measurements of clinic blood pressure without the use of antihypertensive drugs, SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg) Arrhythmia (QT interval prolongation, ventricular tachycardia, ventricular flutter, ventricular fibrillation, frequent ventricular premature beats (24-hour ventricular premature load ≥ 15% of total heart rate), degree atrioventricular block, heart rate<30-40 bpm), congestive heart failure, unstable angina or myocardial infarction, New York Heart Association (NYHA) class II, III, IV heart failure, clinically significant pericardial disease;
11. Participants are known to have chronic obstructive pulmonary disease (COPD) (defined as forced expiratory volume in one second [FEV1]<60% of the predicted normal value), persistent asthma, or a history of asthma within the past 2 years (intermittent asthma or mild persistent asthma allowed to be controlled). Participants with known or suspected COPD must undergo FEV1 testing during the screening period.
12. Patients who undergo major surgeries within 30 days prior to enrollment that significantly reduce their physical condition and increase the risk of thrombosis, or whose surgical plans are scheduled during the study period. Participants who plan to undergo surgical procedures under local anesthesia that will not significantly affect the patient's physical condition and significantly increase the risk of thrombosis formation are eligible to participate in the study;
13. Any clinically significant medical disease or condition that the researcher believes may affect compliance with the experimental protocol or the subject's ability to give informed consent;
14. The subject is a pregnant or lactating female;
15. Uncontrolled hypertension or uncontrolled diabetes;
16. Patients who are allergic to the experimental drug;
17. According to the protocol or the researcher's judgment, patients with serious physical or mental illnesses may interfere with their participation in this clinical study; Drug abuse, medical, psychological, or social conditions that may interfere with subject participation in research or evaluation of research results;
18. Patients undergoing other experimental drug treatments;
19. Participants who have participated in other clinical trials within one month;
20. Any other patients deemed unsuitable for inclusion by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 12 (each cycle is 28 days)
  the rate of very good partial response or better

SECONDARY OUTCOMES:
OS | At the end of Cycle 12 (each cycle is 28 days)
  overall survival
PFS | At the end of Cycle 12 (each cycle is 28 days)
  Progression-free survival
MRD negative rate | At the end of Cycle 12 (each cycle is 28 days)
  the rate of minimal residual disease negativity